CLINICAL TRIAL: NCT00867854
Title: Treatment De-Intensification and Residual HIV-1 in Adolescents and Young Adults: A Sub-Study of ATN 061 and ATN 071.
Brief Title: Treatment De-Intensification and Residual HIV-1 in Youth
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 081
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV-1; HIV Infections
Keywords: de-intensification; HAART; monotherapy; persistent low-level viremia (LLV); treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental: 25 evaluable subjects from the experimental arm of ATN 061 who undergo de-intensification to boosted atazanavir (ATV) with VL suppression of < 100 copies/ml and CD4+ T cells > 350 cells/mm3 at week 48 and maintain VL suppression to < 400 copies/ml with stable CD4+ T cell counts after week 48.
  Interventions: Other: Blood draw
- Control: 25 evaluable subjects from ATN 071 will also be enrolled. These subjects will have initiated HAART according to current DHHS guidelines (CD4+ T cells < 350 cells/mm3), had viral load suppression to < 100 copies/ml at 24 through 48 weeks on HAART and maintained suppression to < 400 copies/ml through week 80.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — This sub-study does not involve additional treatment of any ATN 061 or ATN 071 study subjects. The only intervention involved is the requirement for whole blood collection (40 ml and 60 ml) to be drawn at the same time as four ATN 061 study visits (36, 48, 56, and 80 weeks) for subjects co-enrolled into ATN 061. When these time points coincide with ATN 061 Central Laboratory samples, the 60 ml blood sample will not be collected. For subjects co-enrolled into ATN 071, there are also two samples of whole blood collection (40 ml and 60 ml) required to be drawn at four time points but at weeks 36, 48, 56, and 80 after the initiation of HAART.

SUMMARY:
This laboratory-based sub-study of ATN 061 and ATN 071 will examine the effect of early treatment followed by treatment de-intensification to atazanavir/ritonavir (ATV/r) monotherapy on steady-state frequencies of replication-competent CD4+ T cell Human Immunodeficiency Virus (HIV)-1 reservoirs or cell-associated infectivity (CAI) and persistent low-level viremia (LLV), and their contribution to successful long-term control of HIV-1 replication among HIV-1 infected adolescents and young adults.

ELIGIBILITY:
081 participants must first be enrolled in either ATN 061 or ATN 071 and meet the eligibility criteria of those protocols in addition to those below.

Inclusion Criteria:

061 Participants

* Currently on treatment with an ATV/r-based HAART regimen (ATV/r, FTC, TDF is the preferred regimen);
* HIV-1 viral load < 100 copies at week 24;
* CD4+ T cell count > 350 cells/mm3 at week 24; and
* Able to provide informed consent for the sub-study and adhere to the protocol.

  071 Participants
* Initiated HAART according to current DHHS guidelines (CD4+ T cells < 350 cells/ mm3);
* Currently on treatment with a PI-containing HAART regimen; subjects taking a protease inhibitor OTHER than ATV/r must receive approval by the team via the ATN QNS;
* Plasma HIV-1 viral load < 100 copies at week 24 on HAART; measurement to be collected from clinical care results contained in the medical record at the clinical site within +/- 30 days of week 24 on therapy;
* CD4+ T cell count > 350 cells/mm3 at week 24 on HAART; measurement to be collected from clinical care results contained in the medical record at the clinical site within +/- 30 days of week 24 on therapy; and
* Able to provide informed consent for the sub-study and adhere to the protocol.

General Exclusion Criteria:

* Currently enrolled in the Standard Care Arm of ATN 061;
* Pregnancy or breast feeding;
* Severe (Grade ≥ 3) anemia or other conditions that would not allow adequate blood volume to be drawn;
* Active treatment for systemic infections;
* Treatment with immune modulators, including immunosuppressive or immune modulating therapy (IL-2, intravenous gammaglobulin, and therapeutic or other experimental vaccines including HIV-1 vaccine given for primary prevention at any time (short courses (<14 days) of prednisone for reactive airway disease (RAD) are permitted);
* Active hepatitis B infection as defined by Hepatitis B antigen (Ag) positive;
* Disallowed Medications (see Section 5.3.2);
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with adherence to the study; or
* History of chronic renal insufficiency or Grade 3 or greater serum creatinine.

  061-Specific Exclusion Criteria
* History of an Acquired Immunodeficiency Syndrome (AIDS)-defining illness;
* Meets any ATN 061 exclusion criteria for de-intensification; or
* Meets any ATN 061 premature study discontinuation criteria.

  071-Specific Exclusion Criteria: None

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty-five subjects enrolled in Arm A of ATN 061 who started highly-active antiretroviral therapy (HAART) at CD4+ T cells > 350 cells/cubic millimeter (mm3) and are undergoing treatment de-intensification at week 48 of HAART.
  Twenty-five "control" subjects initiating HAART based on current Department of Health and Human Services (DHHS) guidelines at CD4+ T cell levels < 350 cells/mm3 and maintained on standard HAART.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Steady-state frequencies of replication-competent CD4+ T cell HIV-1 reservoirs in participants starting HAART before DHHS guidelines (CD4+ T cell levels < 350 cells/mm3) vs. those initiating HAART by current DHHS guidelines. | 80 weeks
Quantitative changes in LLV between 6.5 and 50 copies/ml in participants starting early therapy & de-intensifying to ATV/r monotherapy vs. those initiating HAART at CD4+ T cell levels < 350 cells/mm3 & maintaining standard HAART. | 80 weeks
Quantitative changes in viral diversity during HAART in participants initiating early therapy & de-intensifying to ATV/r monotherapy vs those initiating HAART at CD4+ T cell levels < 350 cells/mm3 & maintaining standard HAART. | 80 weeks
Effect of viral diversity in replication-competent CD4+ T cell reservoirs & low viremia variants before de-intensification on successful control of HIV-1 replication during ATV/r maintenance in participants starting HAART before DHHS guidelines. | 80 weeks

SECONDARY OUTCOMES:
To examine the contribution of LLV genotypes, through analysis of the Gag/protease and RT, among subjects who developed rebound viremia above 50 copies/ml during treatment de-intensification to ATV/r. | 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Persaud, M.D., Study Chair — Adolescent Trials Network
Locations (17):
- United States (16):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University - IMPAACT Site, Washington D.C., District of Columbia
  - Children's Diagnostic and Teatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - John Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University - IMPAACT Site, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: ATN website — http://www.atnonline.org